CLINICAL TRIAL: NCT06065891
Title: Prevalence and Consequences of Para-aortic Lymph Node Metastasis in Resectable Pancreatic Cancer: a Prospective Population Based Multicenter Study. The PALN Study
Brief Title: Para-aortic Lymph Node Metastasis in Resectable Pancreatic Cancer
Acronym: PALN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jon Unosson (Other)
Responsible Party: Sponsor-Investigator, Jon Unosson, Principal Investigator, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALN
Record Dates: First submitted 2023-09-08; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pancreas Cancer; Pancreas Adenocarcinoma; Lymph Node Metastasis
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resection of Paraartic lymph nodes (Other): Single arm
  Interventions: Procedure: PALN resection

INTERVENTIONS:
Procedure: PALN resection — Resection of paraaortic lymph nodes in pancreatic cancer

SUMMARY:
Lymph node metastases are a strong prognostic predictor for pancreatic cancer. Para-aortic lymph nodes (PALN) are the final nodes for periampullary cancers before the cancer cells enter the systemic lymphatic circulation. Some consider these nodes to be regional lymph nodes and dissect them as a part of a routine lymphadenectomy for pancreatic cancer. Others argue that metastases to these nodes represent systemic disease and recommend that radical surgery including extended lymphadenectomy should be abandoned.

The aim of this study is to define the incidence and clinical consequences of PALN metastasis in patients submitted to a tentative curative resection for carcinoma of the head of the pancreas by systematically resecting paraaortic lymph nodes.

Primary outcome

1) To determine incidence of PALN metastasis in patients submitted to a tentative curative resection

Secondary outcomes

1. To determine prognosis of patients with PALN metastasis after a curative resection
2. To determine incidence of metastasis in reginal lymph nodes in patients submitted to a tentative curative resection.
3. To determine prognosis of patients with metastasis in regional lymph nodes in patients submitted to a tentative curative resection.
4. To address the question of how to optimize the frozen section analyses of PALN as related to the final pathology report.

300 patients are planned to be included in the trial.

DETAILED DESCRIPTION:
Lymph node metastases are a strong prognostic predictor for pancreatic cancer. Para-aortic lymph nodes (PALN) (No. 16 nodes) are the final nodes for periampullary cancers before the cancer cells enter the systemic lymphatic circulation. Some consider these nodes to be regional lymph nodes and dissect them as a part of a routine lymphadenectomy for pancreatic cancer. Others argue that metastases to these nodes represent systemic disease and recommend that radical surgery including extended lymphadenectomy should be abandoned. There is no consensus whether to abort the resection if metastases in PALN are discovered pre- or perioperatively. Use of adjuvant and neoadjuvant chemotherapy may further affect the impact of lymph node metastases, including PALN.

The aim of this study is to define the incidence and clinical consequences of PALN metastasis in patients submitted to a tentative curative resection for carcinoma of the head of the pancreas by systematically resecting paraaortic lymph nodes.

Primary outcome

1) To determine incidence of PALN metastasis in patients submitted to a tentative curative resection

Secondary outcomes

1. To determine prognosis of patients with PALN metastasis after a curative resection
2. To determine incidence of metastasis in reginal lymph nodes in patients submitted to a tentative curative resection.
3. To determine prognosis of patients with metastasis in regional lymph nodes in patients submitted to a tentative curative resection.
4. To address the question of how to optimize the frozen section analyses of PALN as related to the final pathology report.

PALN are resected separately and analyzed both as cryo sections and by routine histochemistry.

Prevalence of PALN differ markedly from 5% to 30%. Given the descriptive primary endpoint, no rigorous power calculation can be made. Assuming a prevalence of 17% (as reported in a recent series from Stockholm), a hazard ratio for survival ranging from 1,04 to 3,00 and and a drop out of 17%. Complete data is needed for 90 patients but the trial aim to include 300.

Resection of PALN is becoming routine at most participating centers in the trial. Therefore, the trial will not alter care for the participating patients in any major way. Rather the trial aims to systematically asses how this altered practice affect patient outcome.

ELIGIBILITY:
Inclusion Criteria:

Resectable suspected periampullary cancer (requiring duodenopancreatectomy) (NCCN guidelines 2020)

Borderline resectable periampullary cancer (requiring duodenopancreatectomy) (NCCN guidelines 2020)

Age >18 years

Written patient consent

Exclusion Criteria:

Contraindication for a radical resection procedure

Unresectable tumor (NCCN guidelines 2020) or metastatic disease (lgll station 16 not included)

Mental or organic disorders which could interfere with giving informed consent or receiving treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of paraaortic lymph nodes in pancreatic cancer in patients submitted to a tentative curative resection | 5 years
  Frequency of metastases in paraaortic lymph nodes in patients with resectable pancreatic cancer will be assessed by systematically resecting these glands, irrespective of perioperative findings.

SECONDARY OUTCOMES:
To determine prognosis of patients with PALN metastasis (lgll station 16) after a curative resection | 6 years
  Overall survival in years from resection will be measured in patients with and without PALN metastasis
To determine incidence of metastasis in lgll station 8, 9 and 12 in patients submitted to a tentative curative resection. | 5 years
  Frequency of metastases in lymph node 8, 9 and 12 in patients with resectable pancreatic cancer will be assessed by systematically resecting these glands and placing them i separate vials as opposed to en-bloc with the main specimen in order to determine rate of lymph node metastases.
To determine prognosis of patients with metastasis in lgll station 8, 9 and 12 in patients submitted to a tentative curative resection. | 6 years
  Overall survival in years from resection will be measured in patients with and without metastases in lymph node stations 8, 9 and 12.
To address the question of how to optimize the frozen section analyses (lgll station 16) as related to the final pathology report? | 5 years
  Overall survival in years from resection will be measured in patients with and without metastasis in PALN detected on cryosection

CONTACTS AND LOCATIONS:
Overall Officials: Britt-Marie Karlson, Principal Investigator — Uppsala University Hospital
Locations (6):
- Odense University Hospital, Odense, Denmark
- Sweden (5):
  - Sahlgrenska university hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
May be available upon reasonable request